CLINICAL TRIAL: NCT06308393
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial Evaluating the Safety and Pharmacokinetic Profile of RSS0393 Ointment as a Single and Multiple Dose Ascending Local Dermal Administration in Healthy and Adult Subjects With Psoriasis
Brief Title: Randomized, Double-blind, Placebo-controlled Study of RSS0393 Ointment in Healthy and Psoriatic Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSP61418
Record Dates: First submitted 2024-02-05; First posted 2024-03-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Psoriatic Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group 1 (Experimental): Single dose in healthy subjects
  Interventions: Drug: RSS0393 ointment；Placebo
- Treatment group 2 (Experimental): Multiple dose in healthy subjects
  Interventions: Drug: RSS0393 ointment；Placebo
- Treatment group 3 (Experimental): Multiple dose in patients
  Interventions: Drug: RSS0393 ointment；Placebo

INTERVENTIONS:
Drug: RSS0393 ointment；Placebo — RSS0393 ointment；RSS0393 ointment placebo

SUMMARY:
Randomized, double-blind, placebo-controlled study of RSS0393 ointment in healthy and psoriatic subjects

ELIGIBILITY:
Inclusion Criteria:

- Healthy Volunteers：

1. Sign informed consent before the test, fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the requirements of the test plan
2. The age of signing the informed consent must be ≥18 years old and ≤55 years old, male or female
3. Male subjects weighed ≥50 kg, female subjects weighed ≥45 kg, and body mass index (BMI) was in the range of 19.0~26.0 kg/m2

Patients ：

1. The age of signing the informed consent must be ≥18 years old and ≤55 years old, male or female;
2. Male subject ≥50 kg, female subject ≥45 kg, body mass index (BMI) in the range of 19.0~26.0 kg/m2 (including boundary values)
3. At the time of screening and baseline, the clinical diagnosis of psoriasis was at least 6 months
4. During screening, the condition of the subjects was in a stable stage, requiring no new skin lesions, no continuous expansion of original skin lesions, and no obvious features of skin inflammation within 6 months before screening

Exclusion Criteria:

- Healthy Volunteers：

1. The subject has skin conditions that may affect the evaluation of the administration site
2. Patients with severe infection, severe trauma or major surgical operation within 3 months before screening; Patients who plan to undergo surgery during the trial period and within 2 weeks after the end of the trial;
3. Suspected allergy to the investigational drug product or any component of the investigational drug product
4. Persons who have participated in clinical trials of any drug or medical device within 3 months prior to screening, or who are within 5 half-lives of the drug before screening (if the 5 half-lives exceed 3 months); Participants in clinical trials are defined as those who have given informed consent to clinical trials and have used investigational drugs (including placebo) or investigational medical devices;
5. Those who had a history of smoking in the 3 months prior to screening or those who were positive in the screening period;
6. Alcoholics within 3 months prior to screening or those who test positive for alcohol breath test during screening;
7. Those who have a history of drug abuse, drug dependence or positive drug screening during the screening period;
8. Pregnant or lactating women, pregnancy is defined as the female state from pregnancy to termination of pregnancy and the blood β-HCG test is positive during the screening period;

Patients ：

1. Subjects had skin conditions other than psoriasis that could affect the evaluation of the study drug administration site
2. Suspected allergy to the investigational drug product or any component of the investigational drug product;
3. Subjects had a history of any active malignancy or malignancy in the 5 years prior to the screening visit, except skin squamous cell carcinoma or basal cell carcinoma, or cervical cancer in situ, which had resolved after treatment
4. Pre-existing or current clinically significant cardiovascular, liver, neurological, respiratory, blood, gastrointestinal, immune, and kidney diseases or a history of psychiatric disorders that may affect study results or affect drug absorption, distribution, metabolism, and excretion or place subjects at undue risk
5. Participants who had a history of depression and/or were clinically deemed to be at risk of suicide during the screening period and at baseline were excluded
6. Currently has an active tuberculosis infection, or chest radiography indicates the presence of an active tuberculosis infection
7. Those who had undergone any surgery within 1 month prior to screening, or had not recovered as determined by the investigator, or had planned any surgery between the study period and 4 weeks after the study ended
8. The white blood cell count, neutrophil count, lymphocyte count, or hemoglobin in the blood routine examination during screening were out of the normal reference range and were deemed unsuitable for participation in this study by the investigators
9. Screening hepatitis B surface antigen, hepatitis C antibody, HIV antibody test any of the positive results;
10. Individuals who have participated in clinical trials of any drug or medical device within 3 months prior to signing the informed consent or within 5 half-lives of the investigational drug (whichever is older) (except those who have participated in other clinical trials but failed to be screened and administered)
11. The subject has any other condition that the investigator or sponsor considers unsuitable for study participation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The percent of Local skin tolerance was assessed as moderate or higher（Single dose in healthy subjects） | 0.5, 2, 4, 12 post -dose day 1, day 2, day 3, day 5, and day 8
The percent of Local skin tolerance was assessed as moderate or higher （Multiple dose in healthy subjects） | 0.5, 2, 4, 12 post-dose day 1, 0.5post-dose on day2、day3、day4、day5、day6, 0.5, 2, 4, 12 post-dose day7, day8, day9, day11, day14
Measurement of blood examination（Multiple dose in patients ） | Day 1, day 28, day 42 post-dose
Measurement of urine examination（Multiple dose in patients ） | Day 1, day 28, day 42 post-dose
Measurement of Blood Chemistry examination（Multiple dose in patients ） | Day 1, day 28, day 42 post-dose
Measurement of coagulation function examination（Multiple dose in patients ） | Day 1, day 28, day 42 post-dose

SECONDARY OUTCOMES:
AUC0-t （Single dose in healthy subjects） | pre-dose,1, 2 , 4, 8, 12 , 24, 48, 96, 168 post-dose
AUC0-∞（Single dose in healthy subjects） | pre-dose, 1, 2 , 4, 8, 12 , 24, 48, 96, 168 post-dose
Tmax（Single dose in healthy subjects） | pre-dose, 1, 2 , 4, 8, 12 , 24, 48, 96, 168 post-dose
Cmax（Single dose in healthy subjects） | pre-dose, 1, 2 , 4, 8, 12 , 24, 48, 96, 168 post-dose
t1/2（Single dose in healthy subjects） | pre-dose, 1, 2 , 4, 8, 12 , 24, 48, 96, 168 post-dose
CL/F（Single dose in healthy subjects） | pre-dose, 1, 2 , 4, 8, 12 , 24, 48, 96, 168 post-dose
Vz/F（Single dose in healthy subjects） | pre-dose, 1, 2 , 4, 8, 12 , 24, 48, 96, 168 post-dose
AUC0-t （Multiple dose in healthy subjects） | pre-dose, 1 ,2 , 4 , 8 , 12 , 24 post-dose Day1; pre-dose Day5 ; pre-dose Day6; pre-dose Day7; 1 , 2 , 4 , 8 , 12 , 24 , 48 , 96 , 168 post-dose Day7
AUC0-∞（Multiple dose in healthy subjects） | pre-dose, 1 ,2 , 4 , 8 , 12 , 24 post-dose Day1; pre-dose Day5 ; pre-dose Day6; pre-dose Day7; 1 , 2 , 4 , 8 , 12 , 24 , 48 , 96 , 168 post-dose Day7
Tmax（Multiple dose in healthy subjects） | pre-dose, 1 ,2 , 4 , 8 , 12 , 24 post-dose Day1; pre-dose Day5 ; pre-dose Day6; pre-dose Day7; 1 , 2 , 4 , 8 , 12 , 24 , 48 , 96 , 168 post-dose Day7
Cmax（Multiple dose in healthy subjects） | pre-dose, 1 ,2 , 4 , 8 , 12 , 24 post-dose Day1; pre-dose Day5 ; pre-dose Day6; pre-dose Day7; 1 , 2 , 4 , 8 , 12 , 24 , 48 , 96 , 168 post-dose Day7
t1/2（Multiple dose in healthy subjects） | pre-dose, 1 ,2 , 4 , 8 , 12 , 24 post-dose Day1; pre-dose Day5 ; pre-dose Day6; pre-dose Day7; 1 , 2 , 4 , 8 , 12 , 24 , 48 , 96 , 168 post-dose Day7
CL/F（Multiple dose in healthy subjects） | pre-dose, 1 ,2 , 4 , 8 , 12 , 24 post-dose Day1; pre-dose Day5 ; pre-dose Day6; pre-dose Day7; 1 , 2 , 4 , 8 , 12 , 24 , 48 , 96 , 168 post-dose Day7
Vz/F（Multiple dose in healthy subjects） | pre-dose, 1 ,2 , 4 , 8 , 12 , 24 post-dose Day1; pre-dose Day5 ; pre-dose Day6; pre-dose Day7; 1 , 2 , 4 , 8 , 12 , 24 , 48 , 96 , 168 post-dose Day7
Absolute change in PASI score relative to baseline（Multiple dose in patients ） | Day 7, Day 14, Day 28 post-dose
The percentage change in PASI score relative to baseline（（Multiple dose in patients ） | Day 7, Day 14, Day 28 post-dose
The percentage of PASI50、PASI75、PASI90、PASI100（Multiple dose in patients ） | Day 7, Day 14, Day 28 post-dose
The percentage of subjects' achieving PGA score of 0 or 1 and which improvement ≥ 2 from baseline （Multiple dose in patients ） | Day 7, Day 14, Day 28 post-dose
The percentage of subjects' inPGA score improvement ≥ 2 from baseline（Multiple dose in patients ） | Day 7, Day 14, Day 28 post-dose
Absolute change in BSA score relative to baseline（Multiple dose in patients ） | Day 7, Day 14, Day 28 post-dose
The percentage change in BSA score relative to baseline（Multiple dose in patients ） | Day 7, Day 14, Day 28 post-dose
Pharmacokinetics (PK) : Concentrations of RSS0393（Multiple dose in patients ） | Day1 ,Day 7, day 14, Day 28
Pharmacokinetics (PK) : The major metabolites of RSS0393（Multiple dose in patients ） | Day1 ,Day 7, day 14, Day 28

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of University of Science and Technology of China (USTC)., Hefei, Anhui
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided